CLINICAL TRIAL: NCT03687086
Title: A Novel Mechanism for Helping Older Adults Discontinue Use of Sleeping Pills
Brief Title: Sleep Without Insomnia or The Use of Chronic Hypnotics
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Virginia Commonwealth University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Constance Fung, MD, MSHS, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-001009; R01AG057929 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-27 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Medicare Part A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program A (Experimental): cognitive behavioral therapy type A plus medications in packaging type A
  Interventions: Other: Program A
- Program B (Active Comparator): cognitive behavioral therapy type B plus medications in packaging type B
  Interventions: Other: Program B

INTERVENTIONS:
Other: Program A — Cognitive behavioral therapy type A plus medications prepared in packaging type A.
  Arms: Program A
Other: Program B — Cognitive behavioral therapy type B plus medications in packaging type B.
  Arms: Program B

SUMMARY:
Sleeping medications, called hypnotics, are often prescribed for insomnia and are associated with adverse health outcomes in older adults. Response rates to hypnotic discontinuation programs are often inadequate, and many patients eventually resume use of hypnotics, suggesting that other mechanisms need to be targeted to achieve and sustain high rates of non-use. Current programs focus on the tapering of hypnotics and/or the treatment of insomnia symptoms. These programs employ strategies such as supervised gradual taper, cognitive behavioral therapy targeting hypnotic withdrawal, and/or cognitive behavioral therapy for insomnia. Evidence suggests that another mechanism involving "placebo" effects may be a viable target for achieving and sustaining higher discontinuation rates. Cognitive expectancies play a key role in producing placebo effects, which are characterized as real improvements in sleep arising from psychosocial aspects of treatment rather than drug effects alone. In this study, investigators are comparing two programs for discontinuing hypnotic medications-a program that addresses placebo effects associated with hypnotic use and a program that does not address these effects.

DETAILED DESCRIPTION:
Investigators will complete a 5-year randomized trial, recruiting participants from two healthcare systems using a three-step screening process that minimizes time and travel burden to participants. Step 1 (identification of participants): Investigators will identify participants aged >= 55 years who have current prescriptions for lorazepam, temazepam, alprazolam, and/or zolpidem for >= 3 months. Investigators will use three sources to identify these patients: medication lists from electronic health records/administrative data, consults to insomnia clinic, and referrals from providers. The research team will mail a recruitment letter (with opt-out card) to patients identified from these sources. Step 2 (phone screening for current or prior insomnia and current hypnotic use); Patients who endorse a history of insomnia symptoms and current hypnotic use will be invited for an in-person screening. Step 3 (in-person screening for remaining eligibility criteria (and baseline assessments): After written consent, the in-person screening visit consists of a comprehensive sleep, mental health, and brief physical health assessment. Individuals who meet study criteria and agree to continue will be randomized to receive either the Program A (N=94) or Program B (N=94). The interventions are approximately 2 months. Following intention-to-treat principles, all randomized participants will complete an assessment immediately after the intervention ends and 6 months after completing treatment. Participants will be compensated monetarily for assessment visits. Investigators will measure hypnotic expectancies, hypnotic discontinuation, and insomnia severity post-treatment and at 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 55 years
* Use of lorazepam, alprazolam, temazepam,and/or zolpidem for current or prior insomnia symptoms 2 or more nights per week for at least 3 months
* Current or prior insomnia symptoms
* Available to attend weekly in-person sessions over 9 weeks

Exclusion Criteria:

High risk for complications in outpatient hypnotic discontinuation program:

* Seizure disorder
* Supratherapeutic or high baseline hypnotic dose (> diazepam-equivalent of 8 mg/night).
* High baseline risk of complicated withdrawal;benzodiazepine intoxication or current or past symptoms of complicated benzodiazepine/alcohol withdrawal (e.g.,seizure, delirium at baseline (prior to taper))
* Polydrug use (e.g., chronic high dose opioids)
* Unable to keep study medications in secure location
* Evidence of prescription fraud (e.g., multiple prescriptions for same drug filled at multiple pharmacies during overlapping time periods, diversion)

Discontinuation of hypnotic not appropriate:

•Study-targeted hypnotic used to treat another clinical condition (e.g., panic disorder)

Poor candidate for cognitive behavioral therapy for insomnia:

* Presence of bipolar disorder
* Cognitive impairment (e.g., Mini-Mental State Examination < 24)
* Sleep/wake difficulty is better explained by another sleep disorder such as restless legs syndrome, narcolepsy, insufficient sleep syndrome, or circadian rhythm sleep-wake disorders
* Untreated sleep-disordered breathing (respiratory event index >= 15 and < 30 plus excessive daytime sleepiness, or REI >=30)
* Medically/psychiatrically unstable (e.g., planned major surgery during the study period;psychosis, suicidal, active alcohol/substance abuse based on history and medical records)
* Unstable housing situation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Fung, MD, MSHS, Principal Investigator — UCLA, VA Greater Los Angeles
Locations (2):
- United States (2):
  - VA Greater Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
Compliance at one of the sites is not permitting data sharing.

REFERENCES:
- [Derived] Fung CH, Alessi C, Martin JL, Josephson K, Kierlin L, Dzierzewski JM, Moore AA, Badr MS, Zeidler M, Kelly M, Smith JP, Cook IA, Der-Mcleod E, Ghadimi S, Naeem S, Partch L, Guzman A, Grinberg A, Mitchell M. Masked Taper With Behavioral Intervention for Discontinuation of Benzodiazepine Receptor Agonists: A Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1448-1456. doi: 10.1001/jamainternmed.2024.5020. PMID 39374004
- [Derived] Ghadimi S, Grinberg A, Mitchell MN, Alessi C, Moore AA, Martin JL, Dzierzewski JM, Kelly M, Badr MS, Guzman A, Smith JP, Zeidler M, Fung CH. Sleep characteristics and use of multiple benzodiazepine receptor agonists in older adults. J Am Geriatr Soc. 2023 Dec;71(12):3924-3927. doi: 10.1111/jgs.18528. Epub 2023 Aug 1. No abstract available. PMID 37526436

RESULTS

PARTICIPANT FLOW:
Groups:
- Program A: Cognitive Behavioral Therapy for Insomnia, plus novel cognitive and behavioral exercises addressing placebo mechanisms. Medications were prepared in weekly masked blister packs.
  Each participant began the taper with the dose and frequency of the medication that they had been previously prescribed by their provider at the time of the baseline assessment. The taper aimed to reduce the medication by 25% per week over a 9-week period.
- Program B: Cognitive Behavioral Therapy for Insomnia type B plus medications provided in usual form in a standard medication container.
  Each participant began the taper with the dose and frequency of the medication that they had been previously prescribed by their provider at the time of the baseline assessment. The taper aimed to reduce the medication by 25% per week over a 9-week period.
Period: Overall Study
Arm/Group | Program A | Program B
Started | 92 | 96
Completed | 87 | 89
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0
Not completed — Incomplete assessment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Program A | Program B | Total
Number analyzed (Participants) | 92 | 96 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.8) | 69.4 (7.8) | 69.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 61 | 62 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 79 | 89 | 168
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 7 | 17
  White | 72 | 76 | 148
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 92 | 96 | 188
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Mean score on Insomnia Severity Index. This 7-item scale measures self-reported severity of insomnia symptoms. Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
  units on a scale | 13.8 (6.9) | 14.3 (5.7) | 14.0 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Hypnotic Discontinuation
Description: The percentage of participants who had stopped taking a benzodiazepine or z-drug at follow-up. This outcome was measured with 7-day self-reported medication logs.
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Population: For this outcome, the analysis is performed only on those participants who completed the 6-month follow-up assessment and provided data on medication usage. As a result, there were 87 in program A and 89 in program B who met these criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Program A | Program B
Number analyzed (Participants) | 87 | 89
Participants | 64 | 52
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = .039, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.03 to 3.70], Standard Error of Mean 0.63

2. Secondary Outcome: Insomnia Severity Index
Description: Mean score on Insomnia Severity Index. This 7-item scale measures self-reported severity of insomnia symptoms.
  Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
score on a scale | 7.35 (0.58) | 6.47 (0.57)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.155, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (9 Weeks vs. baseline); Mean Difference (Net) = 1.38, 95% CI 2-sided [-0.52 to 3.29], Standard Error of Mean 0.97

3. Secondary Outcome: Insomnia Severity Index
Description: as for outcome 2
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
score on a scale | 7.36 (0.69) | 7.71 (0.68)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.880, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (6 months vs. baseline); Median Difference (Net) = .16, 95% CI 2-sided [-1.88 to 2.20], Standard Error of Mean 1.04

4. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep - Medication Subscale
Description: These 3-items were used to measure hypnotic expectancies. Items ranged from 0 (strongly disagree/least expectancy) to 10 (strongly agree/most expectancy). The scale score is the average of the 3 items and ranged from 0-10 with higher scores indicating greater hypnotic expectancy. Higher hypnotic expectancies are worse outcomes, lower hypnotic expectancies are better outcomes.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
score on a scale | 2.38 (0.25) | 2.72 (0.24)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.228, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (9 weeks vs. baseline); Mean Difference (Net) = -.48, 95% CI 2-sided [-1.25 to 0.30], Standard Error of Mean 0.39

5. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep - Medication Subscale
Description: These 3-items were used to measure hypnotic expectancies. Items ranged from 0 (strongly disagree/least expectancy) to 10 (strongly agree/most expectancy).The scale score is the average of the 3 items and ranged from 0-10 with higher scores indicating greater hypnotic expectancy. Higher hypnotic expectancies are worse outcomes, lower hypnotic expectancies are better outcomes.
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
score on a scale | 3.37 (0.30) | 3.33 (0.30)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.843, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (6 months vs. baseline); Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.96 to 0.78], Standard Error of Mean 0.44

6. Secondary Outcome: Rates of Hypnotic Discontinuation
Description: The percentage of participants who had stopped taking a benzodiazepine or z-drug one week after the end of treatment . This outcome was measured with 7-day self-reported medication logs.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Population: For this outcome, the analysis is performed only on those participants who completed the post-intervention assessment and provided data on medication usage. As a result, there were 86 in program A and 92 in program B who met these criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Program A | Program B
Number analyzed (Participants) | 86 | 92
Participants | 76 | 62
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 3.68, 95% CI 2-sided [1.67 to 8.12], Standard Error of Mean 1.48

7. Secondary Outcome: Hypnotic Dose
Description: The mean daily dose based on self-reported 7-day medication log (in diazepam-equivalent milligrams).
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Measure: Mean (Standard Error); unit: diazepam-equivalent milligrams
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
diazepam-equivalent milligrams | 0.40 (0.16) | 0.57 (0.16)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.443, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (9 weeks vs. baseline); Mean Difference (Net) = -0.32, 95% CI 2-sided [-1.14 to 0.50], Standard Error of Mean 0.42

8. Secondary Outcome: Hypnotic Dose
Description: The mean daily dose based on self-reported 7-day medication log (in diazepam-equivalent milligrams).
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Measure: Mean (Standard Error); unit: diazepam-equivalent milligrams
Arm/Group | Program A | Program B
Number analyzed (Participants) | 92 | 96
diazepam-equivalent milligrams | 1.05 (0.32) | 1.32 (0.32)
Statistical Analysis 1: Comparison: Program A vs Program B; Test type: Superiority; p = 0.409, Mixed Models Analysis; Interaction contrast of Treatment Group (Program A vs. Program B) by Time (6 months vs. baseline); Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.41 to 0.58], Standard Error of Mean 0.51

9. Other Pre Specified Outcome: Digit Symbol Substitution
Description: This test measures processing speed, working memory, visuospatial processing, and attention. It is sensitive to cognitive impairment and change in cognition. The score is based on the number of symbols that the person correctly substitutes in 90 seconds. Total score can range from 0 to 135, with higher scores indicating better cognitive performance.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

10. Other Pre Specified Outcome: Digit Symbol Substitution
Description: as for outcome 9
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

11. Other Pre Specified Outcome: Mini-Mental State Examination
Description: This is a 30-item test of cognitive function. Scores range from 0-30, with higher scores indicating better cognitive function.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

12. Other Pre Specified Outcome: Mini-Mental State Examination
Description: as for outcome 11
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

13. Other Pre Specified Outcome: Trail Making Test A and B
Description: Objective measure of cognitive executive functioning. The scores is the number of seconds it takes to complete the test. Lower scores indicate better cognitive functioning.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

14. Other Pre Specified Outcome: Trail Making Test A and B
Description: as for outcome 13
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

15. Other Pre Specified Outcome: One-leg Balance Test
Description: Objective measure of balance. Participants are timed while they stand on one-leg for up to 60 seconds. Score is the number of seconds able to stand on one-leg. Higher scores indicate better balance.
Time Frame: One week post intervention (which is an average of 9 weeks from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

16. Other Pre Specified Outcome: One-leg Balance Test
Description: as for outcome 15
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Adverse events were collected over approximately 8-months (date of randomization until 6-months after treatment).
Arm/Group | Program A | Program B
All-Cause Mortality (participants affected / at risk) | 1/92 | 0/96
Serious Adverse Events (participants affected / at risk) | 4/92 | 0/96
Other Adverse Events (participants affected / at risk) | 5/92 | 6/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Program A (N=92) | Program B (N=96)
Hospitalization for respiratory viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death from COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Program A (N=92) | Program B (N=96)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gout attack requiring ED visit (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COVID-19 requiring ED visit (Infections and infestations) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Knee pain with torn meniscus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Parasomnia prior to receiving study medication (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was interrupted by the COVID-19 pandemic. Protocol changes were made in response to the COVID-19 pandemic (see protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03687086/Prot_SAP_000.pdf